CLINICAL TRIAL: NCT05839717
Title: Determination of the Clonality Profile in Myeloproliferative Neoplasms and Association With the Thrombotic Complications (CLOJAK)
Acronym: CLOJAK
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/16
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Myeloproliferative Neoplasms; Thrombosis; Clonality; JAK2V617F
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PV and ET patients: The cohort will be composed of PV and ET patients, some with a history of thrombosis and some without any history of thrombosis. A comparison will also be performed between patients with different MPN (PV or ET) and the type of thrombosis (venous, arterial, splanchnic)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — A specific blood sampling will be performed in addition to the classical evaluations that are performed in routine practice

SUMMARY:
Myeloproliferative Neoplasms (MPN) are associated with an increased risk of thrombosis. Platelets, red blood cells (RBC), leukocytes and endothelial cells are involved in these complications. An association with the JAK2V617F allele burden assessed in leukocytes has also been suggested. In some patients the allele burden measured in platelets and red blood cells is higher than the one determined in leukocytes. Our project aims at associating the risk of thrombosis with the allele burden determined in the cell populations (platelets, red blood cells, granulocytes and endothelial cells) and identifying high-risk clonality profiles.

DETAILED DESCRIPTION:
Myeloproliferative Neoplasms (MPN) are hematological malignancies associated with an increased risk of thrombosis. Although different cell types have been involved in these complications (platelets, red blood cells, leucocytes and endothelial cells), there do not exist any reliable biomarker to predict the thrombotic risk in MPN patients. While some studies suggested that the JAK2V617F allele burden measured in leukocytes was associated with the risk of thrombosis, other studies did not confirm these results. Besides, a recent work demonstrated that in some patients, the JAK2V617F allele burden measured in platelets and red blood cells was higher than the one determined in leukocytes. Moreover, some patients present JAK2V617F mutated endothelial cells, known as pro-thrombotic in in vitro and animal models. The CLOJAK project will search for an association between the thrombotic risk in MPN and the proportion of cells carrying the JAK2V617F mutation in erythroid cells and platelets or its presence in endothelial cells. The objective is to determine a clonality profile (i.e. the profile of repartition of the JAK2V617F allele burden in the different hematopoietic and endothelial lineages) associated with the occurrence of thrombosis in MPN patients.

One hundred and twenty PV and ET patients will be studied at diagnosis. Their platelets, red blood cells, granulocytes and endothelial cells will be isolated. The JAK2V617F allele burden will be measured in these cells thanks to a digital PCR technic. An association between the clonality profile and the existence of a thrombosis at diagnosis, the MPN phenotype (PV or ET), the IPSET-thrombosis score and the type of thrombosis (venous, arterial, splanchnic) will be searched.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years)
* Inclusion at diagnosis or during the year following the diagnosis of PV or ET (2016 WHO criteria except bone marrow biopsy that is optional), before introduction of a cytoreductive treatment
* Patient carrying a JAK2V617F mutation
* Subject registered with a social security scheme
* Written informed consent obtained
* Acceptance of inclusion in the FIMBANK registry (specific consent form needed)

Exclusion Criteria:

* ET or PV Patient not carrying a JAK2V617F mutation
* Patient with cytoreductive treatment (hydroxyurea, anagrelide, interferon, ruxolitinib or other chemotherapy) at the time of blood sampling
* Person under judicial safeguards, trustee or curatorship
* Person unable to give her consent
* Non-cooperative person
* Exclusion period after another clinical study or participation to another clinical study in the 30 days before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Myeloproliferative Neoplasms (MPN) carrying a JAK2V617F mutation
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
History of thrombosis at MPN diagnosis | At inclusion
  History of thrombosis at MPN diagnosis defined as the occurrence of a venous (deep vein thrombosis, pulmonary embolism) or arterial thrombosis (ischemic stroke or myocardial infarction) or a thrombosis in the splanchnic area

SECONDARY OUTCOMES:
The JAK2V617F allele burden measured in red blood cells | At inclusion
The JAK2V617F allele burden measured in platelets | At inclusion
The JAK2V617F allele burden measured in granulocytes | At inclusion
The presence of the JAK2V617F mutation in endothelial cells | At inclusion
The clonality profile | At inclusion
  The clonality profile defined based on the association of cell lineages in which a JAK2V617F allele burden over 25% is measured together with the detection (or not) of the JAK2V617F mutation in endothelial cells
The type of MPN according to the 2016 WHO classification of hematological malignancies | At inclusion
The IPSET-Thrombosis score | At inclusion
The type of thrombosis | At inclusion

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU d'Angers, Service Maladies du Sang, Angers
  - CH de Bayonne, Service Hématologie Clinique, Bayonne
  - CHU de Bordeaux, Service Médecine Interne et Maladies Infectieuses, Bordeaux
  - Institut Bergonié, Service Hématologie Clinique, Bordeaux
  - CHU de Brest, Service Hématologie Clinique, Brest
  - CH de Dax, Service Hématologie Clinique, Dax
  - CH de Libourne, Service Hématologie Clinique, Libourne
  - CH de Mont de Marsan, Service Oncologie, Mont-de-Marsan
  - CHU de Bordeaux, Service Hématologie Biologie, Pessac
  - CHU de Bordeaux, Service Hématologie Clinique et Thérapie Cellulaire, Pessac
  - CHU de Bordeaux, Service Médecine Interne, Pessac

IPD SHARING:
Plan to Share IPD: No